CLINICAL TRIAL: NCT01519986
Title: The Effect of Fat on Vitamin D Absorption After a Single Oral Dose
Brief Title: The Effect of Fat on Vitamin D Absorption
Acronym: VITD_100484
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Rio Grande do Sul (Other)
Collaborators: Hospital de Clinicas de Porto Alegre (Other); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Fabiana Viegas Raimundo, Master Degree, Federal University of Rio Grande do Sul
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: VITD_100484
Record Dates: First submitted 2012-01-05; First posted 2012-01-27 (Estimated); Last update posted 2012-01-27 (Estimated); Status verified 2012-01

CONDITIONS: Vitamin D Deficiency
Keywords: Vitamin D; Cholecalciferol; Supplementation; Dietary Supplements; Dietary Fats; 25-hydroxyvitamin D
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Low fat Meal (Experimental): 50,000 UI vitamin D3 with low fat meal
  Interventions: Dietary Supplement: Vitamin D3; Dietary Supplement: Placebo
- Medium fat meal (Experimental): 50,000 UI vitamin D3 with medium fat meal
  Interventions: Dietary Supplement: Vitamin D3; Dietary Supplement: Placebo
- High fat meal (Experimental): 50,000 UI vitamin D3 with high fat meal
  Interventions: Dietary Supplement: Vitamin D3; Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin D3 — Supplement of vitamin D3
Dietary Supplement: Placebo — Placebo

SUMMARY:
The purpose of this study is to evaluate the absorption of dietary supplement of vitamin D3 (cholecalciferol), through the variation of 25 (OH) D levels, as the fat content of the meal associated with the administration of the supplement.

ELIGIBILITY:
Inclusion Criteria:

Residents of the hospital clinics of Porto Alegre

Exclusion Criteria:

* Don't drink milk
* Obesity
* Malnutrition
* Liver disease
* Kidney disease or diabetes
* Use of dietary supplements containing calcium and vitamin D
* Medications
* Anticonvulsants
* Barbiturates, or steroids.
* Having performed a journey the last four months to locations near the Earth's equatorial plane, due to sun exposure that may have occurred during this period, or vacations planned during the study period.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2011-09; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline in serum 25(OH)D at 14 day after intervention | Change from baseline in serum 25(OH)D at 14 days
  25(OH)D response to supplemental vitamin D3

SECONDARY OUTCOMES:
Change from baseline in Parathyroid hormone at 14 days after intervention | Change from baseline in Parathyroid hormone at 14 days
  Parathyroid hormone response to supplemental vitamin D3

CONTACTS AND LOCATIONS:
Overall Officials: Tania W Furlanetto, PhD, Principal Investigator — Federal University of Health Science of Porto Alegre; Gustavo AM Faulhaber, PhD, Study Chair — Federal University of Health Science of Porto Alegre; Fabiana V Raimundo, MD, Study Chair — Federal University of Health Science of Porto Alegre

REFERENCES:
- [Background] Raimundo FV, Faulhaber GA, Menegatti PK, Marques Lda S, Furlanetto TW. Effect of High- versus Low-Fat Meal on Serum 25-Hydroxyvitamin D Levels after a Single Oral Dose of Vitamin D: A Single-Blind, Parallel, Randomized Trial. Int J Endocrinol. 2011;2011:809069. doi: 10.1155/2011/809069. Epub 2011 Dec 7. PMID 22190928
- [Background] Avnur Z, Nathan I, Dvilansky A, Livne A. Plasma constituent (s) inhibiting platelet adhesiveness. Isr J Med Sci. 1977 Mar;13(3):264-71. PMID 15956